CLINICAL TRIAL: NCT00817999
Title: The Impact of Grapefruit Juice on the Response to a Loading Dose and Maintenance Dose of Clopidogrel in Healthy Volunteers
Brief Title: The Impact of Grapefruit Juice on the Response to Clopidogrel
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: 08-15073
Record Dates: First submitted 2009-01-06; First posted 2009-01-07 (Estimated); Results first posted 2012-10-01 (Estimated); Last update posted 2012-10-01 (Estimated); Status verified 2012-08

CONDITIONS: Healthy
Keywords: Platelet Aggregation Inhibition
MeSH Terms: interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Loading Dose (Experimental): Participants received a 300 mg dose of clopidogrel with or without GFJ.
  Interventions: Dietary Supplement: Grapefruit juice; Drug: Clopidogrel 300 mg
- Maintenance Dose (Experimental): Participants received clopidogrel 75 mg/day for 7 days with or without GFJ
  Interventions: Dietary Supplement: Grapefruit juice; Drug: Clopidogrel 75 mg/day

INTERVENTIONS:
Dietary Supplement: Grapefruit juice — Participants received grapefruit juice during 1 of the 2 periods.
Drug: Clopidogrel 75 mg/day
  Arms: Maintenance Dose
Drug: Clopidogrel 300 mg
  Arms: Loading Dose

SUMMARY:
This study will measure the percentage of platelet aggregation inhibition with a loading dose of clopidogrel (300 mg) using the VerifyNow Assay System in healthy volunteers who have drank 11 oz of grapefruit juice. It will also measure the percentage of platelet aggregation inhibition with a maintenance dose of clopidogrel (75 mg/day) using the VerifyNow Assay System in healthy volunteers who have drank 11 oz grapefruit juice daily.

DETAILED DESCRIPTION:
This study will examine the effect of GFJ on the loading dose (300 mg) of clopidogrel and will evaluate the effect of GFJ on the maintenance dose (75 mg/day) of clopidogrel. Subjects will be randomized to either initially receive GFJ prior to their loading dose of clopidogrel or receive GFJ prior to their second loading dose. The subjects who have been randomized to receive GFJ initially will drink two small cans (11 oz total) of regular strength GFJ in the morning, followed two hours later by a loading dose (300 mg) of clopidogrel and will then return to the clinic 6 hours after their loading dose to have their platelet inhibition measured. Subjects will have ~ 5 milliliters (1 teaspoonful) of whole blood drawn from an antecubital vein in their forearm via a 21 gauge needle attached to a blue-top plastic vacuette sodium citrate blood collection (Greiner, Monroe, NC) tube to test inhibition of platelet aggregation. After their first loading dose, a 2 week washout period will follow to allow for their platelet aggregation to return to normal. Following the washout period, the subjects will take their second loading dose of clopidogrel and again return to the clinic for platelet inhibition measurement. The same timing will be followed for the loading dose taken without prior GFJ.

During the maintenance dose phase of this study, subjects will take 75 mg/day clopidogrel for 7 days with or without GFJ. Subjects will be randomized to either GFJ during the first period or GFJ during the second period. A minimum 2 week washout period will occur between the two 7 day courses of clopidogrel. Platelet inhibition measurement will occur at the end of each 7 day period as described above.

ELIGIBILITY:
Inclusion Criteria:

* Ages 19-40
* Health status confirmed by medical history and physical examination and laboratory analysis

Exclusion Criteria:

* Pregnancy
* Taking routine prescription or over-the-counter prescriptions
* Taken over-the-counter analgesic/anti-inflammatory medication within two weeks of study participation
* Recently had grapefruit juice or regularly drinks grapefruit juice

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2008-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tammy Burns, PharmD, Principal Investigator — Creighton Cardiac Center
Locations (1):
- Creighton Cardiac Center, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Loading Dose: Healthy volunteers who received a 300 mg dose of clopidogrel with or without grapefruit juice.
- Maintenance Dose: Healthy volunteers who received clopidogrel 75 mg/day for 7 days during each period with or without grapefruit juice.
Period: Grapefruit Juice
Arm/Group | Loading Dose | Maintenance Dose
Started | 15 | 17
Completed | 15 | 17
Not Completed | 0 | 0
Period: No Grapefruit Juice
Arm/Group | Loading Dose | Maintenance Dose
Started | 15 | 17
Completed | 15 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Loading Dose | Maintenance Dose | Total
Number analyzed (Participants) | 15 | 17 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 17 | 32
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 24.4 (5.9) | 25.47 (5.66) | 25.47 (5.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 23
  Male | 5 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United States | 15 | 17 | 32

OUTCOME MEASURES:

1. Primary Outcome: % Platelet Inhibition
Description: % platelet inhibition measured by Verify Now
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: percentage of platelet inhibition
Arm/Group | Loading Dose With Grapefruit Juice | Maintenance Dose With Grapefruit Juice | Loading Dose Without Grapefruit Juice | Maintenance Dose Without Grapefruit Juice
Number analyzed (Participants) | 15 | 17 | 15 | 17
percentage of platelet inhibition | 23.4 (14.2) | 24.6 (24.2) | 41.2 (19.1) | 59 (22.5)

ADVERSE EVENTS:
Arm/Group | Loading Dose | Maintenance Dose
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/17
Other Adverse Events (participants affected / at risk) | 0/15 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes